CLINICAL TRIAL: NCT01381562
Title: A Study to Assess the Safety, Tolerability and Preliminary Efficacy of GSK2251052 in the Treatment of Complicated Intra-abdominal Infection in Adults
Brief Title: GSK2251052 in the Treatment of Complicated Intra-abdominal Infections
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Microbiological findings of resistance on therapy in patients with complicated urinary tract infection
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114689
Record Dates: First submitted 2011-06-09; First posted 2011-06-27 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Infections, Intestinal
Keywords: intra-abdominal infection; belly; Gram-negative pathogen; abscess; peritonitis
MeSH Terms: conditions — Infections; Intraabdominal Infections; Abscess; Peritonitis | interventions — 3-(aminomethyl)-7-(3-hydroxypropoxy)-1-hydroxy-1,3-dihydro-2,1-benzoxaborole; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GSK2251052 750mg (Experimental): q12h administered via IV infusion, plus saline placebo
  Interventions: Drug: Drug: GSK2251052; Other: Placebo
- GSK2251052 1500mg (Experimental): q12h administered via IV infusion, plus saline placebo
  Interventions: Drug: Drug: GSK2251052; Other: Placebo
- Meropenem 1G (Active Comparator): q8h administered via IV infusion, plus saline placebo
  Interventions: Drug: Meropenem; Other: Placebo

INTERVENTIONS:
Drug: Drug: GSK2251052 — Reconstituted, added to 250mL 0.9% NaCl solution and administered via IV infusion
  Arms: GSK2251052 1500mg; GSK2251052 750mg
Drug: Meropenem — Reconstituted, added to 100mL 0.9% NaCl solution and administered via IV infusion
  Other Names: Merrem ®; Meronem
  Arms: Meropenem 1G
Other: Placebo — saline placebo

SUMMARY:
This study is being conducted to evaluate the safety, efficacy and pharmacokinetics/pharmacodynamics of GSK2251052 in subjects with complicated intra abdominal infections. GSK2251052 will be compared to meropenem, an IV therapy that is approved for use in the treatment of subjects with cIAI. GSK2251052 has a spectrum of microbiological activity that includes pathogens responsible for cIAI.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects least 18 years of age.

N.B. Females of non-childbearing or childbearing potential may be enrolled. It is not contraindicated to enrol females of childbearing potential; however, females of childbearing potential must have a negative pregnancy test at study entry and must have practiced adequate contraception for at least 30 days prior to study entry. Additionally, the subject agrees to one of the following methods for avoidance of pregnancy during the entire study treatment period:

* Abstinence; or,
* Oral Contraceptive, either combined estrogen/progesterone or progesterone alone, PLUS an additional barrier method [ie, condom, occlusive cap (diaphragm or cervical/vault caps) or vaginal spermicidal agent (foam/gel/film/cream/suppository)]; or,
* Injectable progesterone; or
* Implants of levonorgestrel; or,
* Estrogenic vaginal ring; or,
* Percutaneous contraceptive patches; or
* Intrauterine device (IUD) or intrauterine system (IUS) showing that failure rate is less than 1% in the IUD or IUS product label; or,
* Has a male partner who is sterilized (vasectomy with documentation of azoospermia).
* Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Females are considered to be of non-childbearing potential if they have documented tubal ligation or hysterectomy; or are postmenopausal, defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]
* Subject has evidence of a systemic inflammatory response believed to be related to an intra-abdominal infectious process with no evidence of another infectious source (e.g., catheter related, lung, urinary tract)
* Subject has an abnormal white blood cell count (>12,000/µL or <4,000/µL or >10% bands) PLUS one or more of the following
* Fever, defined as >38°C oral, >38.5°C tympanic or >39°C rectal, within the last 24 hours
* Heart rate of more than 90 beats per minute
* Respiratory rate of more than 20 breaths per minute or a PaCO2 level of less than 32 mm Hg
* Altered mental status thought due to an infectious process
* Subject is post-op and required surgery within the last 24 hours prior to first dose of study medication OR subject requires surgical intervention (e.g., laparotomy, laparoscopic surgery, or percutaneous drainage of an abscess) within 24 hours of first dose of study medication with no more than one pre-surgical dose of an antibiotic given for pre-operative prophylaxis.
* Subject has a known Gram-negative pathogen(s) isolated prior to study entry or a suspected Gram-negative post-operative infection or has failed a prior Gram negative treatment regimen

A subject enrolled as a failure of a previous antibacterial treatment regimen must:

Show lack of improvement or worsening in signs and symptoms of infection, including continued or worsening peritoneal findings Require additional surgical intervention which must be performed within 24 hours of first dose of study medication with no more than one pre-surgical dose of an antibiotic given for pre-operative prophylaxis AND/OR Be post-op and have required surgery within 24 hours prior to first dose of study medication with no more than one pre-surgical dose of an antibiotic given for pre-operative prophylaxis.

Have a culture positive for a Gram-negative pathogen (from an intra-abdominal site) N.B. Such subjects may be enrolled before the results of the culture are known but if the culture is negative, the subject must be removed from study drug therapy.

* Subject requires antibacterial therapy for an anticipated duration of 7 days or more, in addition to surgical intervention, for one of the following eligible diagnoses:
* Cholecystitis (including gangrenous cholecystitis) with rupture, perforation or progression of the infection beyond the gallbladder wall
* Diverticular disease with perforation or abscess
* Appendiceal perforation with duration of symptoms >=48 hours AND imaging that is strongly suggestive of free fluid or abscess
* Acute gastric and duodenal perforations, only if operated more than 24 hours after perforation occurred
* Traumatic perforation of the intestine only if operated more than 12 hours after perforation occurred
* Peritonitis due to perforated viscus, post-operative, or other focus of infection (but not spontaneous bacterial peritonitis associated with cirrhosis and chronic ascites)
* Inflammatory bowel disease or ischemic bowel disease with bowel perforation
* If pre-operative, subject must have peritoneal findings highly suspicious for cIAI, defined as one or more of the following:
* Abdominal pain and/or tenderness
* Localized or diffuse abdominal wall rigidity
* An imaging procedure, ie. ultrasound or CT scan showing evidence of IAI
* Mass
* Ileus
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block

Exclusion Criteria:

* Subject has a known or suspected diagnosis of the following:
* Abdominal wall abscess
* Small bowel obstruction or ischemic bowel disease without perforation
* Traumatic bowel perforation with surgery within 12 hours
* Perforation of gastroduodenal ulcer with surgery within 24 hours
* Any other intra-abdominal processes in which the primary etiology is not likely to be infectious.
* Simple cholecystitis
* Gangrenous or suppurative cholecystitis without rupture or extension beyond the gallbladder wall
* Simple appendicitis
* Acute suppurative cholangitis
* Infected, necrotizing pancreatitis, or pancreatic abscess
* Subject must not be managed by staged abdominal repair or open abdominal technique
* Subject is known at study entry, prior to randomization to study medication, to have a cIAI caused by a Gram-positive pathogen or a pathogen resistant to the study antimicrobial agent.
* Subject has an APACHE II score >20.
* Subject is considered unlikely to survive the 4 6 week study period or has any rapidly progressing disease or immediately life-threatening illness (including acute hepatic failure, respiratory failure or septic shock).
* Subject requires treatment with concomitant systemic antibacterial agents other than vancomycin.
* Subject has moderate to severe impairment of renal function including a calculated creatinine clearance (CrCl) of less than 50 mL/min; requirement for peritoneal dialysis, hemodialysis, or hemofiltration; or oliguria (less than 20 mL urine output per hour over 24 hours).
* Subject has a prior history of seizures or CNS abnormality and/or is using concomitant medications with seizure potential
* Subject requires probenecid or valproic acid medications
* Subject has evidence of known or pre-existing severe hepatic disease(Child-Pugh score of B or C)
* Subject has a known baseline hemoglobin less than 10 g/dL ,hematocrit less than 30% and/or a known reticulocyte count of >5% (ie, reticulocytes >5% of total RBC mass)
* Subject has known neutropenia or is anticipated to develop neutropenia during the course of the study (ie, new chemotherapy patient), with absolute neutrophil count less than 1000 cells/mm3
* Subject has a known platelet count less than 75,000 cells /mm3 (subjects with platelet counts as low as 50,000 cells /mm3 are eligible if the reduction is historically stable)
* Subject has an immunocompromising illness; including known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), organ (including bone marrow) transplant recipients, and hematological malignancy, and immunosuppressive therapy , including high-dose corticosteroids (e.g., greater than 40mg prednisone or equivalent per day for greater than two weeks)
* Subject has participated in any investigational drug or device study within 30 days of study entry or within 5 half-lives, whichever is longer.
* Subject has had more than 24 hours of systemic antibacterial therapy for cIAI within the 48 hour period prior to first dose of IV study drug therapy, unless there is a documented lack of clinical response to such therapy
* Subject has a history of moderate or severe hypersensitivity to Meropenem or to beta-lactam antibiotics
* Subject has previously received treatment with GSK2251052
* Subject is pregnant or nursing.
* Subject, in the opinion of the investigator, may be significantly compromised by a potential drop in haemoglobin greater than 2.5g/dl which is not related to the condition under study
* French subjects: the French subject has participated in any study using an investigational drug during the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-10-03 (Actual); Primary Completion 2012-03-05 (Actual); Study Completion 2012-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (29):
- United States (12):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Lima, Ohio
  - GSK Investigational Site, Richmond, Virginia
- Canada (4):
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
- GSK Investigational Site, Prague, Czechia
- France (3):
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Strasbourg
- GSK Investigational Site, Verona, Veneto, Italy
- Russia (4):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburgh
  - GSK Investigational Site, Smolensk
- Spain (4):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pama de Mallorca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at five centers in four countries (United Stated of America, Spain, France and Russia) between 03-October-2011 and 05-March-2012.
Pre-assignment Details: A total of 15 participants were enrolled in the study; of those, 5 participants each were randomised to receive GSK2251052, 750 milligram (mg) or 1500 mg or meropenem 1.0 gram (g), intravenously. One participant in the GSK2251052 1500 mg group was randomised but not treated, thus safety and efficacy populations consisted of 14 participants.
Groups:
- GSK2251052 750 mg: Eligible participants received GSK2251052, 750 mg, in 200 or 250 millilitre (mL) saline solution as intravenous (IV) infusion administered over 60 minutes, twice a day (BID) and meropenem matching placebo solution, 100 ml, administered over 30 minutes, thrice a day (TID) from Day 2 to Day 14 of the study.
- GSK2251052 1500 mg: Eligible participants received GSK2251052, 1500 mg, in 200 or 250 mL saline solution as IV infusion administered over 60 minutes, BID and meropenem placebo solution, 100 ml, administered over 30 minutes, TID from Day 2 to Day 14 of the study.
- Meropenem 1.0 g: Eligible participants received meropenem, 1.0 g, in 100 ml saline solution as IV infusion administered over 30 minutes TID and two doses of GSK2251052 matching placebo saline solution, 200 or 250 ml, administered over 60 minutes, BID from Day 2 to Day 14 of the study.
Period: Overall Study
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1.0 g
Started | 5 | 4 | 5
Completed | 5 | 3 | 5
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK2251052 750 mg: Eligible participants received GSK2251052, 750 mg, in 200 or 250 mL saline solution as IV infusion administered over 60 minutes, BID and meropenem matching placebo solution, 100 ml, administered over 30 minutes, TID from Day 2 to Day 14 of the study.
- Meropenem 1 g: Eligible participants received meropenem, 1.0 g, in 100 ml saline solution as IV infusion administered over 30 minutes TID and two doses of GSK2251052 matching placebo saline solution, 200 or 250 ml, administered over 60 minutes, BID from Day 2 to Day 14 of the study.
- Total: Total of all reporting groups
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1 g | Total
Number analyzed (Participants) | 5 | 4 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.0 (15.05) | 41.3 (13.65) | 34.6 (10.31) | 36.3 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 4 | 3 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1 | 0 | 1 | 2
  Asian - Central/South Asian Heritage | 0 | 0 | 1 | 1
  Asian - East Asian Heritage | 0 | 1 | 0 | 1
  White - White/Caucasian/European | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE included AEs those result in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition
Time Frame: Up to Day 42
Population: Safety Population comprised of all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Meropenem 1g: Eligible participants received meropenem, 1.0 g, in 100 ml saline solution as IV infusion administered over 30 minutes TID and two doses of GSK2251052 matching placebo saline solution, 200 or 250 ml, administered over 60 minutes, BID from Day 2 to Day 14 of the study.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 5 | 4 | 5
Participants
  Any AE | 5 | 4 | 3
  Any SAE | 2 | 3 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Trends in Vital Signs Over the Period of Study Duration
Description: Vital parameters including systolic and diastolic blood pressure, heart rate, respiration rate, and temperature were recorded. The number of participants with potentially clinically concern value of any vital parameter at any visit were reported.
Time Frame: Up to Day 42
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 5 | 4 | 5
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Normal and Abnormal ECG Findings
Description: 12-lead ECGs was obtained during the study using an ECG machine and performed with the participant in a semi-supine position rested in this position for at least 10 minutes beforehand. Measurements deviated substantially from previous readings were repeated immediately. Number of participants with normal and abnormal ECG findings were reported.
Time Frame: Up to Day 42
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 5 | 4 | 5
Participants
  Baseline, Pre-dose 1, Normal | 4 | 4 | 4
  Baseline, Pre-dose 1, Unable to evaluate | 0 | 0 | 1
  Baseline, Pre-dose 1, Abnormal | 1 | 0 | 0
  Baseline, Pre-dose 2, Normal | 4 | 4 | 5
  Baseline, Pre-dose 2, Abnormal | 1 | 0 | 0
  Baseline, Pre-dose 3, Normal | 4 | 4 | 5
  Baseline, Pre-dose 3, Abnormal | 1 | 0 | 0
  Baseline, Post-dose , Normal | 4 | 3 | 4
  Baseline, Post-dose , Abnormal | 1 | 1 | 1
  On IV Therapy (Day 4), Pre-dose, Normal | 4 | 4 | 5
  On IV Therapy (Day 4), Pre-dose, Abnormal | 1 | 0 | 0
  On IV Therapy (Day 4), Post-dose, Normal | 5 | 4 | 5
  Early Follow-up | 5 | 3 | 5

4. Primary Outcome: Laboratory Parameters of Interest- Mean Hemoglobin Over the Period of Study Duration
Description: Absolute mean hemoglobin values recorded over the period of duration were reported.
Time Frame: Up to Day 42
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Gram per Litre
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 5 | 4 | 5
Gram per Litre
  Baseline (Day 1) | 142.2 (8.76) | 121.5 (12.23) | 125.0 (14.85)
  On IV Therapy (Day 3): number analyzed (Participants) | 5 | 4 | 4
  On IV Therapy (Day 3) | 134.4 (13.61) | 112.3 (16.30) | 137.3 (19.64)
  On IV Therapy (Day 5): number analyzed (Participants) | 5 | 3 | 5
  On IV Therapy (Day 5) | 127.2 (14.79) | 120.7 (11.02) | 131.0 (18.63)
  On IV Therapy (Day 8): number analyzed (Participants) | 1 | 1 | 1
  On IV Therapy (Day 8) | 148.0 (NA) — Only one participant was analyzed. | 132.0 (NA) — Only one participant was analyzed. | 143.0 (NA) — Only one participant was analyzed.
  On IV Therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  On IV Therapy (Day 11) | 97.0 (NA) — Only one participant was analyzed. |  |
  End Of IV Therapy | 126.2 (23.35) | 123.8 (9.88) | 130.8 (20.22)
  Haematology Safety | 131.4 (15.21) | 118.0 (9.93) | 138.6 (14.72)
  Test of cure: number analyzed (Participants) | 4 | 4 | 5
  Test of cure | 131.0 (25.26) | 116.0 (5.77) | 138.2 (11.52)
  Early Follow up: number analyzed (Participants) | 4 | 2 | 4
  Early Follow up | 125.5 (31.16) | 121.5 (3.54) | 138.5 (10.54)
  Late Follow up: number analyzed (Participants) | 5 | 2 | 5
  Late Follow up | 133.2 (19.38) | 126.5 (0.71) | 146.8 (17.25)

5. Primary Outcome: Laboratory Parameters of Interest- Mean Reticulocytes Over the Period of Study Duration
Description: Absolute mean reticulocytes values recorded over the period of duration were reported.
Time Frame: Up to 42 days
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Trillion cells per Litre
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 5 | 4 | 5
Trillion cells per Litre
  Baseline (Day 1) | 0.0589 (0.01839) | 0.0573 (0.00761) | 0.0810 (0.02547)
  On IV Therapy (Day 3): number analyzed (Participants) | 5 | 4 | 4
  On IV Therapy (Day 3) | 0.0487 (0.01874) | 0.0638 (0.03074) | 0.0725 (0.02418)
  On IV Therapy (Day 5): number analyzed (Participants) | 5 | 3 | 5
  On IV Therapy (Day 5) | 0.0580 (0.02377) | 0.0480 (0.00515) | 0.0870 (0.02888)
  On IV Therapy (Day 8): number analyzed (Participants) | 1 | 1 | 1
  On IV Therapy (Day 8) | 0.0077 (NA) — Only one participant was analyzed. | 0.0444 (NA) — Only one participant was analyzed. | 0.0650 (NA) — Only one participant was analyzed.
  On IV Therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  On IV Therapy (Day 11) | 0.0335 (NA) — Only one participant was analyzed. |  |
  End Of IV Therapy | 0.0564 (0.02919) | 0.0602 (0.01899) | 0.0872 (0.02792)
  Haematology Safety | 0.0640 (0.02406) | 0.0478 (0.01937) | 0.0815 (0.03405)
  Test Of Cure: number analyzed (Participants) | 4 | 4 | 5
  Test Of Cure | 0.0959 (0.01260) | 0.0860 (0.01764) | 0.0846 (0.01270)
  Early Follow up: number analyzed (Participants) | 5 | 2 | 4
  Early Follow up | 0.0842 (0.02559) | 0.0769 (0.00537) | 0.0796 (0.02874)
  Late Follow up: number analyzed (Participants) | 5 | 2 | 5
  Late Follow up | 0.1046 (0.02945) | 0.0870 (0.01018) | 0.0828 (0.01431)

6. Primary Outcome: Mean Change From Baseline in Hemoglobin for Partcipants With Significant Hemoglobin Drop
Description: Participants in whom the hemoglobin level dropped by more than 30% from Baseline that was not attributable to acute blood loss were recorded and immediately withdrawn from study treatment. Baseline assessments were recorded on Visit 1 (Day 1) and used as Baseline values. The change from Baseline was calculated by subtracting the Baseline values from Day 42 values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing. The mean change from Baseline in hemoglobin for participants with significant hemoglobin drop were reported.
Time Frame: Baseline (Day 1) and up to Day 42
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: grams/L
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 5 | 4 | 5
grams/L
  On IV Therapy, Day 3: number analyzed (Participants) | 5 | 3 | 2
  On IV Therapy, Day 3 | -7.8 (18.07) | -13.3 (8.62) | 0.0 (9.90)
  On IV Therapy, Day 5: number analyzed (Participants) | 5 | 2 | 3
  On IV Therapy, Day 5 | -15.0 (18.88) | 1.5 (3.54) | -1.7 (8.62)
  On IV Therapy, Day 8: number analyzed (Participants) | 1 | 1 | 0
  On IV Therapy, Day 8 | 3.0 (NA) — Only one participants was available at the time of analysis. Dispersion was not calculated. | -6.0 (NA) — Only one participants was available at the time of analysis. Dispersion was not calculated. |
  On IV Therapy, Day 11: number analyzed (Participants) | 1 | 0 | 0
  On IV Therapy, Day 11 | -58.0 (NA) — Only one participants was available at the time of analysis. Dispersion was not calculated. |  |
  End of IV Therapy: number analyzed (Participants) | 5 | 3 | 3
  End of IV Therapy | -16.0 (28.88) | -0.7 (3.79) | -2.3 (3.79)
  Hematology Safety: number analyzed (Participants) | 5 | 3 | 3
  Hematology Safety | -10.8 (22.48) | -8.3 (13.80) | 10.0 (8.72)
  Test for Cure: number analyzed (Participants) | 4 | 3 | 3
  Test for Cure | -13.3 (32.09) | -8.7 (15.95) | 11.0 (10.58)
  Early Follow-up: number analyzed (Participants) | 4 | 2 | 2
  Early Follow-up | -16.5 (39.31) | 6.0 (5.66) | 1.5 (7.78)
  Late Follow-up: number analyzed (Participants) | 5 | 2 | 3
  Late Follow-up | -9.0 (25.82) | 11.0 (9.90) | 20.0 (2.65)

7. Primary Outcome: Number of Participants With Clinical Response at Test of Cure Visit (5-9 Days Post-therapy) in Microbiological Intent to Treat (MITT) Population
Description: Test of cure-clinical success was resolution of signs and symptoms of complicated intra-abdominal infection (cIAI) for participants who were clinical successes at the end of IV therapy visit with no new symptoms recorded that were not present at Baseline and no use of additional antibiotic therapy for cIAI. Test of cure-clinical failure was persistence of signs and symptoms of cIAI recorded at Baseline, or reappearance of signs and symptoms that had previously resolved, or new signs and symptoms recorded that were not present at a previous visit, or receipt of additional or alternate antibiotic therapy for cIAI or participant had died. Test of cure- unable to determine was refusal to consent to a clinical examination, lost to follow-up. Participants who were 'unable to determine' at End of IV therapy were considered 'unable to determine' Test of cure Visit as well. Due to early termination of the study, a Bayesian approach for informal hypothesis testing was not performed.
Time Frame: Day 5 to 9 post IV therapy
Population: MITT Population comprised of all randomized participants who received at least one dose of study medication and had at least one Gram-negative pathogen identified at Baseline. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 4 | 2 | 4
Participants
  Test of Cure Clinical Success | 3 | 1 | 4
  Test of Cure Clinical Failure | 1 | 1 | 0

8. Secondary Outcome: Number of Participants With Clinical Response at Test of Cure Visit (5-9 Days Post-therapy) in Microbiological Evaluable Population.
Description: as for outcome 7
Time Frame: Day 5 to 9 post IV therapy
Population: Microbial evaluation population comprised of participants from the MITT population who adhered to the protocol (do not violate the protocol) and received at least 5 days of IV therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 4 | 2 | 4
Participants
  Test of Cure Clinical Success | 3 | 1 | 4
  End of IV Clinical Failure | 1 | 1 | 0

9. Secondary Outcome: Number of Participants With Microbiological Response in MITT Population
Description: Microbiological Response at End of IV Therapy was assessed as Microbiological Success (MS) or Microbiological Failure (MF). MS was categorized as microbiological eradication (ME) and presumed microbiological eradication (PME). MF was categorized as microbiological persistence (MP), presumed microbiological persistence (PMP), unable to determine, new infection and colonization. Number of participants with microbiological response in MITT population were reported.
Time Frame: End of IV therapy (0-24 hours post-therapy); Test of cure (5-9 days post-therapy); Late Follow-up (21-28 days post-therapy)
Population: MITT Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 4 | 2 | 4
Participants
  End of IV Therapy, MS, PME | 3 | 1 | 4
  End of IV Therapy, MF, MP | 0 | 1 | 0
  End of IV Therapy, MF, PMP | 1 | 0 | 0
  Test of Cure, MS, PME | 3 | 1 | 4
  Test of Cure, MF, PMP | 1 | 1 | 0
  Late follow-up, MS, PME | 3 | 1 | 4
  Late follow-up, MF, PMP | 1 | 1 | 0

10. Secondary Outcome: Number of Participants With Microbiological Response in Microbiological Evaluable Population
Description: Microbiological Response at End of IV Therapy was assessed as MS or MF. MS was categorized as ME and PME. MF was categorized as MP and PMP, unable to determine, new infection and colonization. Number of participants with microbiological response in microbiological evaluable population were reported.
Time Frame: as for outcome 9
Population: Microbiological evaluable population. Only those participants available at the specified time points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 4 | 2 | 4
Participants
  End of IV Therapy, MS, PME | 3 | 1 | 4
  End of IV Therapy, MF, MP | 0 | 1 | 0
  End of IV Therapy, MF, PMP | 1 | 0 | 0
  Test of Cure, MS, PME | 3 | 1 | 4
  Test of Cure, MF, PMP | 1 | 1 | 0
  Late follow-up, MS, PME | 3 | 1 | 4
  Late follow-up, MF, PMP | 1 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinical Response in Microbiological Evaluable Population
Description: Clinical success was defined as resolution or improvement of Baseline signs and symptoms of cIAI, including white blood cell count within normal limits, participant was afebrile and peritoneal findings consistent with cIAI were no longer present with no new symptoms present that were not present at Baseline and no use of additional or alternate antibiotic therapy. Clinical failure was defined as (1) Lack of improvement or worsening in one or more signs and symptoms of cIAI recorded at Baseline, or reappearance of signs and symptoms that had previously resolved, or (2) signs and symptoms recorded that were not present at Baseline, or (3) receipt of additional or alternate antibiotic therapy for cIAI or (4) participant had died, or (5) participant had an adverse event leading to study drug discontinuation and the participant required additional or alternative antibacterial therapy for the current cIAI.
Time Frame: as for outcome 9
Population: Microbiological evaluable population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 4 | 2 | 4
Participants
  End of IV Therapy, Clinical Success | 3 | 1 | 4
  End of IV Therapy, Clinical Failure | 1 | 1 | 0
  Late follow-up, Follow-up Clinical Success | 3 | 1 | 4
  Late follow-up, End of IV Clinical Failure | 1 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinical Response in MITT Population
Description: as for outcome 11
Time Frame: End of IV therapy (0-24 hours post-therapy) and Late Follow-up (21-28 days post-therapy)
Population: MITT Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 4 | 2 | 4
Participants
  End of IV Therapy, Clinical Success, | 3 | 1 | 4
  End of IV Therapy, Clinical Failure | 1 | 1 | 0
  Late follow-up, Follow-up Clinical Success | 3 | 1 | 4
  Late follow-up, End of IV Clinical Failure | 1 | 1 | 0

13. Secondary Outcome: Number of Participants With Therapeutic Response in Microbiological Evaluable Population
Description: Therapeutic response was a measure of the overall efficacy response, and a therapeutic success referred to participants who had been deemed both a 'clinical success' and a 'microbiological success'. All other combinations (other than 'clinical success' + 'microbiological success') were deemed failures for therapeutic response. Therapeutic response was determined programmatically.
Time Frame: as for outcome 9
Population: Microbiological evaluable population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 4 | 2 | 4
Participants
  End of IV Therapy, Therapeutic Success | 3 | 1 | 4
  End of IV Therapy, Therapeutic Failure | 1 | 1 | 0
  Test of Cure, Therapeutic Success | 3 | 1 | 4
  Test of Cure, Therapeutic Failure | 1 | 1 | 0
  Late Follow-up, Therapeutic Success | 3 | 1 | 4
  Late Follow-up, Therapeutic Failure | 1 | 1 | 0

14. Secondary Outcome: Number of Participants With Therapeutic Response in MITT Population
Description: as for outcome 13
Time Frame: as for outcome 9
Population: MITT Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
Number analyzed (Participants) | 4 | 2 | 4
Participants
  End of IV Therapy, Therapeutic Success | 3 | 1 | 4
  End of IV Therapy, Therapeutic Failure | 1 | 1 | 0
  Test of Cure, Therapeutic Success | 3 | 1 | 4
  Test of Cure, Therapeutic Failure | 1 | 1 | 0
  Late Follow-up, Therapeutic Success | 3 | 1 | 4
  Late Follow-up, Therapeutic Failure | 1 | 1 | 0

15. Secondary Outcome: Maximum Plasma Concentration (Cmax) of GSK2251052
Description: Cmax was planned to be determined. A nonlinear mixed effects model as implemented in the program NONMEM was planned to be used to analyze plasma concentration data. However, data for pharmacokinetics (PK) analysis was not collected.
Time Frame: Day 3: Pre- dose (just prior to the start of the first infusion of the day) and 1 hour (just prior to the end of the infusion), 2, 4, and 12 hours post-dose
Population: PK population consisted of participants for whom PK samples were collected. Data for PK analysis was not collected.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Area Under the Concentration Time Curve (AUC) of GSK2251052
Description: AUC was planned to be determined. A nonlinear mixed effects model as implemented in the program NONMEM was planned to be used to analyze plasma concentration data. However, data for PK analysis was not collected.
Time Frame: as for outcome 15
Population: PK population. Data for PK analysis was not collected.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Time to Cmax (Tmax) of GSK2251052
Description: Tmax was planned to be determined. A nonlinear mixed effects model as implemented in the program NONMEM was planned to be used to analyze plasma concentration data. However, data for PK analysis was not collected.
Time Frame: as for outcome 15
Population: PK population. Data for PK analysis was not collected.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Cmax of GSK2251052 Using Non-intensive PK Sampling
Description: Cmax was planned to be determined. A nonlinear mixed effects model as implemented in the program NONMEM was planned to be used to analyze plasma concentration data. However, data for PK analysis was not collected.
Time Frame: Day 5: Pre- dose (just prior to the start of the first infusion of the day) and 1 hour (just prior to the end of the infusion), 2, 4, and 12 hours post-dose
Population: PK population. Data for PK analysis was not collected.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: AUC of GSK2251052 Using Non-intensive PK Sampling
Description: as for outcome 16
Time Frame: as for outcome 18
Population: PK population. Data for PK analysis was not collected.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Tmax of GSK2251052 Using Non-intensive PK Sampling
Description: as for outcome 17
Time Frame: as for outcome 18
Population: PK population. Data for PK analysis was not collected.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Cmax of GSK2251052 Using Intensive PK Sampling
Description: as for outcome 18
Time Frame: Day 5: Pre-dose (just prior to the start of the first infusion of the day) 0.5, 1 hour (just prior to the end of the infusion), 1.25, 1.5, 2, 3, 4, 8 and 12 hours post-dose
Population: PK population. Data for PK analysis was not collected.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: AUC of GSK2251052 Using Intensive PK Sampling
Description: as for outcome 16
Time Frame: as for outcome 21
Population: PK population. Data for PK analysis was not collected.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Tmax of GSK2251052 Using Intensive PK Sampling
Description: as for outcome 17
Time Frame: as for outcome 21
Population: PK population. Data for PK analysis was not collected.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were reported up to Late Follow-up visit (Day 42)
Description: Safety population was used to used to collect the AEs.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Meropenem 1g
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5 | 3/4 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 4/4 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2251052 750 mg (N=5) | GSK2251052 1500 mg (N=4) | Meropenem 1g (N=5)
Abdominal abscess (Infections and infestations) | 0 | 2 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2251052 750 mg (N=5) | GSK2251052 1500 mg (N=4) | Meropenem 1g (N=5)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1
Infusion site pain (General disorders) | 0 | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 1
Reticulocyte count increased (Investigations) | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Dyssomnia (Psychiatric disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Anisocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Poikilocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early because only 15 participants were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.